CLINICAL TRIAL: NCT02105506
Title: Safety and Feasibility of TachoSil®: Application on Esophageal Anastomoses
Acronym: SAFE-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R. van Hillegersberg (Other)
Responsible Party: Sponsor-Investigator, R. van Hillegersberg, Prof. R. van Hillegersberg, surgeon, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL38212
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Esophageal Disease; Gastric Disease
Keywords: Esophagus; Stomach; Resection; Esophageal disease requiring surgery; Gastric disease requiring surgery
MeSH Terms: conditions — Esophageal Diseases; Stomach Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tachosil patch (Experimental): Tachosil patch (9.5 x 4.8 cm), containing human fibrinogen (5.5 mg/cm2) and human thrombin (2.0 IU/cm2), applied during surgery. Up to 7 patches per participant may be applied.
  Interventions: Drug: Tachosil patch

INTERVENTIONS:
Drug: Tachosil patch

SUMMARY:
Rationale: The construction of esophageal anastomoses is associated with considerable risk at postoperative anastomotic leakage. Application of TachoSil®, a tissue sealant with human fibrinogen and thrombin, can improve strength of the esophageal anastomosis and potentially prevent anastomotic leakage.

Objective: Evaluation of feasibility and safety of TachoSil® application on esophageal anastomoses.

Study design: Non-randomized, non-blinded, single-center intervention study. Study population: Patients, 18-80 years old, undergoing an elective total gastrectomy with an esophago-jejunostomy or esophagectomy with a planned esophagogastric anastomosis will be enrolled. A total number of 15 patients will be included in the study.

Intervention: Gastric or esophageal resection will be executed according to the common procedures used in the UMC Utrecht. After construction of the esophageal anastomosis, all enrolled participants will receive a TachoSil® patch, which will be applied on the esophageal anastomosis intra-operatively. Hence, TachoSil® is used as an add-on therapy. TachoSil® will be degraded enzymatically in a period of approximately 24 weeks after application.

Main study parameters/endpoints: The primary endpoint is feasibility, which is assessed by evaluation of adherence of the patch. A time-action analysis of the application of the Tachosil patch will be performed.

Nature and extent of the burden associated with participation: The burden for the patient is minimal. The total surgical procedure will be prolonged with 10-15 minutes. Postoperative care and outpatient visits do not differ from regular protocol. TachoSil® is approved and registered for supportive treatment in surgery for improvement of haemostasis and to promote tissue sealing by the European Commission.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an elective total gastrectomy with an esophago-jejunostomy or esophagectomy with a planned esophagogastric anastomosis
* Male and female gender
* Ages 18-80
* Signed informed consent
* For females of childbearing potential:

  * Patient uses a reliable contraceptive method: contraceptive pill, intrauterine device, subdermal implantation, or transdermal patch
  * Patient has a negative serum or urine pregnancy test.

Exclusion Criteria:

* Emergency resections of esophagus of stomach
* Unsigned informed consent
* History of hypersensitivity reactions to human fibrinogen, human thrombin, or collagen.
* Patients having difficulty understanding Dutch and English
* Mentally incapable patients
* Pregnancy or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Feasibility | Surgical procedure
  The adherence of the Tachosil patch

SECONDARY OUTCOMES:
all cause mortality | within the first 30 days (plus or minus 3 days) after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands